CLINICAL TRIAL: NCT06395805
Title: Evaluation of Quality of Life and Self-assurance and Social Support Earned in Patients Before and After Operation for Non-cellular Head Cancer and Cancer in the First, Second and Third Stages of Advance
Brief Title: Evaluation of Quality of Life and Self-assurance and Social Support Earned for Non-cellular Head Cancer
Status: Recruiting | Type: Observational
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Edyta Laska, Principal Investigator, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: 31/2023
Record Dates: First submitted 2024-01-01; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Head Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BREF, ADL, AIS. — 1. abbreviated version of the quality of life assessment questionnaire - The World Health Organization Quality of Life (WHOQOL) -BREF
  2. scale I - ADL according to Lawton
  3. the AIS questionnaire
  4. the Zimet Multidimensional Scale of Perceived Social Support - the original version of the MSPSS

SUMMARY:
Research objectives:

* To evaluate the quality of life of patients before and after surgery for benign head tumors ( meningiomas) and malignant tumors at stage I, II and III, to assess whether it depends on the size of the tumor, type of tumor, malignancy and its location
* evaluation of the independence of patients before and after surgery for head tumors at different stages of the disease - benign tumors (meningiomas) and malignant tumors in stage I, II and III, evaluation of what factors affected the different independence of patients
* Multidimensional evaluation of perceived social support of patients before and after surgery for head cancers - benign ( meningiomas) and malignant tumors in stage I, II and III, taking into account three sources of support: significant person, family and friends

Scientific (research) problems:

- What is the quality of life of patients before and after surgery for benign ( meningiomas) and malignant head cancers at stages I, II and III ? Is quality of life in patients with head cancer dependent on tumor size, malignancy, location or type of cancer ?

ELIGIBILITY:
Inclusion criteria for the study:

-clinical diagnosis of head cancer

Study exclusion criteria:

- cranio-brain injuries and inflammatory brain diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each patient who is admitted to the surgical ward with a diagnosis of head cancer will be qualified for surgery will be given written consent for the study and the processing of personal data, as well as information for the researcher with questionnaires, and then give written consent will be recruited for the study. The patient's personal data processing information will be retained for the study until its completion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed using The World Health Organization Quality of Life (WHOQOL) scale. Social support assessed using Zimet's Multidimensional Perceived Social Support Scale. Patient self-efficacy as assessed by the Lawton I-ADL scale and AIS scale. | 12 months to 24 months
  Quality of life assessed using The World Health Organization Quality of Life (WHOQOL-BREF) scale questionnaire which contains 26 questions analyzing four domains of life and separately perception of quality of life and self-assessment of health status.
  It is used to assess the quality of life of both healthy and sick people in clinical practice and addresses the following domains of quality of life: somatic functioning, psychological functioning, social functioning and community functioning.
  Social support assessed using Zimet's Multidimensional Perceived Social Support Scale - the original version on the MSPSS.
  Patients' self-efficacy assessed by the I-ADL scale according to Lawton, where the patient answers nine questions regarding activities of daily living. Disease acceptance scale according to the AIS questionnaire, where the patient answers eight questions regarding their disease.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Raphael's Hospital, Krakow, Lesserpoland, Poland